CLINICAL TRIAL: NCT05145088
Title: Association Analysis of Aerobic Capacity and Expiratory Forced Vital Capacity in Overweight and Obese Adults After Submaximal Exercise Training of Three Weeks (a Randomized Controlled Trial Study)
Brief Title: Association Analysis of Aerobic Capacity and Expiratory Forced Vital Capacity in Overweight and Obese Adults After Submaximal Exercise Training of Three Weeks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FUI/CTR/2021/3
Record Dates: First submitted 2021-11-03; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Overweight and Obese Adults
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are randomly allocated by coin toss method in two groups and they are unawre of random allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The participants in this group are under control and not perfoming any exercise, and their life style is NOT consistent with any kind of submaximal exercise training designed as per protocol.
- Experimental group (Experimental): the particpants are made to perform submaximal exercise testing according to ACSM guidelines for 03 weeks.
  For Moderate-intensity exercises includes either 30 min a day for five days a week or a total of two hours and 30 min per week using 50% to 70% of maximum heart rate.
  The data will be calculated at two times in the form of pre and post testing.
  Interventions: Behavioral: submaximal exercise testing according to ACSM guidelines

INTERVENTIONS:
Behavioral: submaximal exercise testing according to ACSM guidelines — For Moderate-intensity exercises includes either 30 min a day for five days a week or a total of two hours and 30 min per week using 50% to 70% of maximum heart rate
  Arms: Experimental group

SUMMARY:
It is a randomized controlled trial. The study is initiated after getting an approval from ERC FUI. The research is being conducted according to ethical guidelines of Pakistan Medical Research Council and declaration of Helsinki. Confidentiality and anonymity of participants is being maintained throughout the research project. Study subjects are being selected on the basis of inclusion and exclusion criteria and then are being randomly allocated on the basis of coin toss method in Control and experimental groups. An informed consent is being taken from study participants prior to recruiting in study. After random allocation the participants are being given self-administered PAR-Q followed by pre exercise Expiratory forced vital capacity and VO2 max measurements through Digital spirometer and McArdle Katch test respectively. Then study participants will be made to perform submaximal exercise testing according to ACSM guidelines for 03 weeks. The data will be collected at two time intervals that is on day 1 and then after 03 weeks. Data will then be analyzed using SPSS version 21.0.

DETAILED DESCRIPTION:
Objectives of study:

1. To find out association between aerobic capacity and expiratory forced vital capacity in overweight obese adults after submaximal exercise training of 03 weeks.
2. To find out effectiveness of submaximal exercise training of 03 weeks on aerobic capacity and expiratory forced vital capacity in overweight obese adults.

STUDY HYPOTHESIS

Alternate hypothesis: There is a significant association between aerobic capacity and expiratory forced vital capacity in overweight obese adults Null hypothesis: There is no significant association between aerobic capacity and expiratory forced vital capacity in overweight obese adults MATERIAL & METHODS

STUDY DESIGN: Randomized control trial SETTING: FUIRS clinical lab DURATION OF STUDY: 1.5 years SAMPLE SIZE: N=30 (sample size validated through tool)

SAMPLING TECHNIQUE: Non probability convenient sampling

Outcome Measures:

Data will be collected on Demographics and general information. VO2 max is being assessed with the help of McArdle Katch test. FVC is being assesed with the help of hand held spirometer device.

Experimental Group (A) = 03 weeks of submaximal exercise according to ACSM guidelines.

Control group (B) =this group is under control with no exercise training.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study within the community.

An informed consent is being taken from study participants prior to recruiting in study. After random allocation the participants are being given self-administered PAR-Q followed by pre exercise Expiratory forced vital capacity and VO2 max measurement by the PI.

Significance of study:

This study will make people become aware of their current physical fitness level, so the lifestyle behaviors can be modified if needed, in order to improve their quality of life This study will open new doors for researchers to do long term studies by using different parametes of lungs function test available in hand held spirometer.

ELIGIBILITY:
Inclusion criteria:

1. Young adults between age 18 to 35 years
2. Classified Overweight and obese adults according to their BMI

Exclusion criteria:

1. Any prior history of chronic respiratory illness and chronic cardiac disease.
2. Individuals belonging to certain occupations like coal miners, hard rock miners, tunnel workers, concrete manufacturing workers and non-mining industrial workers.
3. Individuals with any diagnosed musculoskeletal disorder.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
VO2 max | Day 1
  It is going to measure the aerobic capacity of the individuals.
VO2 max | 3rd week
  It is going to measure the aerobic capacity of the individuals.

SECONDARY OUTCOMES:
BMI | Day 1
  Change in BMI after submaximal exercise training
BMI | 3rd week
  Change in BMI after submaximal exercise training of 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Summyia Siddique Malik, MSPT, Principal Investigator — Foundation University Islamabad; Dr Sanna Pervaiz, MSPT, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No